CLINICAL TRIAL: NCT04681924
Title: Effects of Low Carbohydrate Diet Compared to Low Fat Diet in Reversing the Metabolic Syndrome Using NCEP ATP III Criteria; Randomized Clinical Trial
Brief Title: Low Carbohydrate Diet Versus Low Fat Diet in Reversing the Metabolic Syndrome Using NCEP ATP III Criteria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Sherzad Ali Ismael, Assistant Professor Dr. Sherzad Ali Ismael, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6122342016
Record Dates: First submitted 2020-10-12; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Low carbohydrate diet group received low carbohydrate food versus low fat diet group who received low fat food. Eight hundred adults (≥18year old) of both gender (358 males and 442 females) are surveyed in the 12 population clusters in Erbil city to estimate the prevalence of MetS. The population frame of household of Erbil population based on all 12 offices of Family ID card in Erbil city. The randomized cluster sampling survey method of the houses is used for sample selection. Out of 289 obese adult participants who had the inclusion criteria to participate in the study, only 94 of them agreed to participate in the intervention (23 males and 71 females). Those 94 are randomly assigned into two groups, the LCD (n=54) and LFD (n=40) group. All the adult participants are completed a comprehensive medical examination and routine blood tests
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low carb diet (Experimental): Low carb diet (n=54)
  Interventions: Other: Diet intervention
- Low fat diet (Experimental): Low fat diet (n=40)
  Interventions: Other: Diet intervention

INTERVENTIONS:
Other: Diet intervention — Low carb diet group are compared to low fat diet group and followed up for 6 months
  Other Names: LCD vs LFD

SUMMARY:
The National Cholesterol Education Program Adult Treatment Panel-III (NCEP ATP III) definition of metabolic syndrome (MetS)is one of the most widely used criteria of metabolic syndrome. It incorporates the key features of hyperglycemia/insulin resistance, visceral obesity, dyslipidemia and hypertension. According to the NCEP ATP III guidelines, in our study, the participants having the metabolic syndrome if they possess three or more of the following criteria: abdominal obesity: Increased waist circumference, Elevated serum triglycerides, Reduced high density lipoprotein cholesterol (HDL), Elevated blood pressure both systolic blood pressure (SBP) and diastolic and Elevated fasting blood glucose.

Although the pathogenesis of MetS is strongly linked to excessive food consumption, in particular fat intake, still there is no consensus about the effects of low carbohydrate diet (LCD) versus low fat diet (LFD) on reversing the MetS and on its metabolic risk factors. However, concerns have been raised with regard to the macronutrient shift with high carbohydrate restriction and the substantial intakes of fats, which may present unfavorable effects on cardiovascular disease risk factors. Meanwhile the LFD has generally been supported by studies to have beneficial effects on these risk factors.

There is no consensus about the effects of LCD versus LFD on the metabolic syndrome. This study investigated the effects of LCD versus LFD on the obese peoples and followed up them for 6 months. Out of 289 obese adults apparently healthy were randomly chosen by a stratified multistage probability sampling method, 94 of them are agreed to participate in the study. They were assigned randomly into low carbohydrate and low-fat diet groups. Both groups were followed up for 6 months and the data were taken at baseline, after 3 months and 6 months of intervention. Ninety-four obese participants completed the intervention.

DETAILED DESCRIPTION:
The metabolic syndrome (MetS) is a major and escalating public health and clinical challenge worldwide in the wake of urbanization, excess energy intake, increasing obesity, and sedentary life style. Metabolic syndrome a five-fold increasing the risk of type 2 diabetes mellitus (T2DM) and two fold increasing the risk of developing cardiovascular disease (CVD) over the next 5 to 10 years. Worldwide prevalence of MetS ranges from <10% to as much as 84%, depending on the region, urban or rural environment, population composition (sex, age, race, and ethnicity), and the definition of the syndrome used. The NCEP ATP III definition is one of the most widely used criteria of metabolic syndrome. It incorporates the key features of hyperglycaemia/insulin resistance, visceral obesity, dyslipidaemia and hypertension.

The treatment of metabolic syndrome intends to improve insulin sensitivity and correct the associated metabolic and cardiovascular abnormalities. During the past few years, several studies have evaluated the health effects of low carbohydrate-high protein diet (LCD), with emphasis on cardiovascular diseases versus low fat diet (LFD). Low-carbohydrate diet has become a popular strategy for weight loss and weight management in recent years. In addition, data from several randomized trials have demonstrated that LCD produced greater effects on weight loss and reducing cardiovascular and metabolic risk factors than LFD. A popular version of this LCD recommends extreme restriction of carbohydrate intake to less than 20 gram/day initially.

Although the pathogenesis of MetS is strongly linked to excessive food consumption, in particular fat intake, still there is no consensus about the effects of LCD versus LFD on reversing the MetS and on its metabolic risk factors. However, concerns have been raised with regard to the macronutrient shift with high CHO restriction and the substantial intakes of fats, which may present unfavorable effects on CVD risk factors. Meanwhile the LFD has generally been supported by studies to have beneficial effects on these risk factors.

The purpose of this study was to investigate the effects of a low carb diet compared to low fat diet on reversing and treating metabolic syndrome and their risk factors among a sample of obese adults in Erbil city/ Iraq Kurdistan.

This study is a randomized clinical trial conducted over 6 months, between (January and June 2017) with outcome assessments at baseline, at 3, and 6 months of intervention.

Eight hundred adults (≥18year old) of both gender (358 males and 442 females) are surveyed in the 12 population clusters in Erbil city to estimate the prevalence of MetS. The population frame of household of Erbil population based on all 12 offices of Family ID card in Erbil city. The randomized cluster sampling survey method of the houses is used for sample selection. Out of 289 obese adult participants who had the inclusion criteria to participate in the study, only 94 of them agreed to participate in the intervention (23 males and 71 females). Those 94 are randomly assigned into two groups, the LCD (n=54) and LFD (n=40) group. All the adult participants are completed a comprehensive medical examination and routine blood tests.

A modified questionnaire of world health organization (WHO) STEPwise approach to Surveillance of noncommunicable diseases (STEPS) was used in this study. The modified questionnaire included 25 questions on socio-demographic (9 questions), anthropometric measurements (7 questions) and biochemical measurements (9 questions).

According to the NCEP ATP III guidelines, in our study, the participants having the metabolic syndrome if they possess three or more of the following criteria is written in the following: Abdominal obesity: Increased waist circumference Men: > 102 cm, Women: > 88 cm, Elevated triglycerides > 150 mg/dL, Reduced HDL Men: < 40 mg/dL, Women: < 50 mg/dL, Elevated blood pressure > 130/85 mm Hg & Elevated fasting glucose > 100 mg/dL.

Individuals with history or diagnosed with diseases and health related issues like diabetes mellitus, hypertension, chronic skin disease, heart disease, hyperlipidemia, malignant disease, and rheumatoid arthritis and those who had undergone surgery during one month before the study are excluded in the study.

More than half of the participants (n = 54) were followed the LCD. In this diet program, the primary behavioral target was to limit carbohydrate intake. Therefore, the limited carbohydrate intake and unrestricted consumption of fat and protein are allowed. During the first two weeks of the intervention, participants were instructed to limit carbohydrate intake to 20-gram per day. After the first two weeks, the participants were instructed to gradually increase 5-gram of the carbohydrate intake every week.

Forty participants were followed the LFD. The primary behavioral target was to limit the overall energy intake (1200 kcal/d). They received instructions to increase calorie intake from 1200 to 1800 kcal per day (≤ 30% of calories from fat, <7% saturated fat).

All 94 participants completed the 6 months of intervention. They were followed up regularly by direct interview every two weeks by the researcher. Each follow-up session lasted 15 to 30 minutes. All of them were prescribed the same level of instruction concerning drinking 10-12 glasses of water /day and physical activity (principally walking), beginning at week 2, with 1 session of 30-45 minutes per day then increasing the duration of physical activity to reach at least 60 minutes /day.

An electronic weight scale (model 770: Seca, Germany) was used to measure the participants' weight to the nearest 0.1 kg. While the participants were asked to stand still without shoes, a measuring tape was utilized to measure their lightly clothed height to the nearest 0.5 cm. The formula used for calculating body mass index (BMI) was as following: BMI=weight(kg)/height(m2). The measurements were collected at baseline, at 3 months and 6 months.

Waist circumference (WC) was measured midway above umbilical between the distal border of the lowest rib and the superior border of the iliac crest at the end of a normal expiration. Measurements were done with the subject in upright position, without clothes, both feet touching the ground, and arms hanging freely. A non-elastic tape measure was placed directly on the skin on the waist line without putting pressure on the abdominal wall.

Blood pressure (BP) was measured by the researcher using an MDF Desk Mercury Sphygmomanometer (Model No: MDF 800), with cuff sizes based on measured arm circumference. Blood pressure checked after participants were asked to sit and take rest for 10 minutes. The measurements were collected at baseline, at 12 and 24 weeks.

Blood samples were obtained after participants fasted overnight (8-10 hours). Blood sample analyzed in the laboratory department of one of the two main hospitals in Erbil city, the Rzgary Teaching Hospital. The serum analyzed by the same laboratory and by the same device (BIOTECNICA BT4500 Full Automated Chemistry Analyser, 2016).

The adherence of the diet programs was done based on participants' self-reporting. Also, delivery of the intervention and assessment of the outcomes are not blinded.

Data on baseline characteristics of adult participants were expressed as means ± SD and/ or frequencies and percentage. The data checked for normal distribution by Shapiro-Wilk test; the p-value was 0.10 which indicates that the data was normally distributed. The study used t tests and Chi square test of association to compare baseline characteristics between both diet programs. When the expected count more than 20% of the cells of the table was less than 5, Fisher exact test was used. An independent samples t-test was used to compare the means of a normally distributed metabolic risk factors for both independent diet programs at the baseline and after 6 months of intervention. A two-way repeated measures ANOVA was used to compare differences of metabolic dependent variables between the two independent variables, the LCD & LFD, at baseline, after 3 months and after 6 months. To determine how much of an effect of intervention has had on the participants, the study used the following cut-offs to interpret the results: 0.14 or more are large effects, 0.06 are medium effects and 0.01 are small effects. A p-value of ≤0.05 was considered as the level of significance for all analyses. The Statistical Package for the Social Sciences (SPSS) software, version 22 was used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

1. All adult obese participants
2. Had 3 or more of the following criteria of metabolic syndrome according to the NCEP

ATP III guidelines:

* Abdominal obesity: increased waist circumference
* Elevated triglycerides
* Reduced HDL
* Elevated blood pressure
* Elevated fasting glucose

Exclusion Criteria:

1. Individuals with history or diagnosed with diseases and health related issues like:

   * Diabetes mellitus
   * Hypertension
   * Chronic skin disease
   * Heart disease
   * Hyperlipidemia
   * Malignant disease
   * Rheumatoid arthritis
2. Those who had undergone surgery during one month before the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-07-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of metabolic syndrome | Baseline
  The number of participants in the sample with the criteria of metabolic syndrome, divided by the total number of participants in the sample.
  According to the NCEP ATP III guidelines, the participants having the metabolic syndrome if they possess three or more of the following criteria: Abdominal obesity, elevated triglycerides, reduced HDL, elevated blood pressure and elevated fasting glucose.
Change from baseline in metabolic syndrome and at 6 months | 6 months
  Data on baseline characteristics of adult participants were expressed as means ± SD and/ or frequencies and percentage. The data checked for normal distribution by Shapiro-Wilk test; the p-value was 0.10 which indicates that the data was normally distributed. The study used t tests and Chi square test of association to compare baseline characteristics between both diet programs. An independent samples t-test was used to compare the means of a normally distributed metabolic risk factors for both independent diet programs at the baseline and after 6 months of intervention.
Compare prevalence of metabolic syndrome in both diet programs | 6 months
  A two-way repeated measures ANOVA was used to compare differences of metabolic dependent variables between the two independent variables, the LCD & LFD, at baseline, after 3 months and after 6 months. To determine how much of an effect of intervention has had on the participants, the study used the following cut-offs to interpret the results: 0.14 or more are large effects, 0.06 are medium effects and 0.01 are small effects.

SECONDARY OUTCOMES:
Body mass index | Baseline
  The formula used for calculating body mass index (BMI) was as following: BMI=weight(kg)/height(m2)
Change from baseline in abdominal obesity and at 6 months | 6 months
  Waist circumference in cm was measured midway above umbilical. Abdominal obesity by increased waist circumference (in men: >= 102 cm while in women: >= 88 cm).
Change from baseline in elevated triglycerides and at 6 months | 6 months
  Blood samples for lipid profile as as mg/ dL were obtained after participants fasted overnight (8-10 hours). The serum analyzed by the(BIOTECNICA BT4500 Full Automated Chemistry Analyser, 2016). Elevated triglycerides if it was >= 150 mg/dL).
Change from baseline in reduced HDL and at 6 months | 6 months
  Blood samples for lipid profile as as mg/ dL were obtained after participants fasted overnight (8-10 hours). The serum analyzed by the(BIOTECNICA BT4500 Full Automated Chemistry Analyser, 2016). Reduced HDL if it was in men: < 40 mg/dL while in women: < 50 mg/dL).
Change from baseline in elevated blood pressure and at 6 months | 6 months
  Blood pressure as mmHg was measured using an MDF Desk Mercury Sphygmomanometer (Model No:MDF 800). elevated blood pressure if it was >= 130/85 mm Hg.
Change from baseline in elevated fasting glucose and at 6 months | 6 months
  Blood samples for blood glucose as as mg/ dL were obtained after participants fasted overnight (8-10 hours). The serum analyzed by the(BIOTECNICA BT4500 Full Automated Chemistry Analyser, 2016).Elevated fasting glucose if it was >= 100 mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Ali A Al-Dabbagh, Prof., Study Director — Hawler Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alberti KG, Eckel RH, Grundy SM, Zimmet PZ, Cleeman JI, Donato KA, Fruchart JC, James WP, Loria CM, Smith SC Jr; International Diabetes Federation Task Force on Epidemiology and Prevention; Hational Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; International Association for the Study of Obesity. Harmonizing the metabolic syndrome: a joint interim statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation; International Atherosclerosis Society; and International Association for the Study of Obesity. Circulation. 2009 Oct 20;120(16):1640-5. doi: 10.1161/CIRCULATIONAHA.109.192644. Epub 2009 Oct 5. PMID 19805654
- [Background] Kaur J. A comprehensive review on metabolic syndrome. Cardiol Res Pract. 2014;2014:943162. doi: 10.1155/2014/943162. Epub 2014 Mar 11. PMID 24711954 (Retraction: PMID 30993018 Cardiol Res Pract. 2019 Jan 31;2019:4301528)
- [Background] Huang PL. A comprehensive definition for metabolic syndrome. Dis Model Mech. 2009 May-Jun;2(5-6):231-7. doi: 10.1242/dmm.001180. PMID 19407331
- [Background] Riccardi G, Rivellese AA. Dietary treatment of the metabolic syndrome--the optimal diet. Br J Nutr. 2000 Mar;83 Suppl 1:S143-8. doi: 10.1017/s0007114500001082. PMID 10889805
- [Background] Gardner CD, Kiazand A, Alhassan S, Kim S, Stafford RS, Balise RR, Kraemer HC, King AC. Comparison of the Atkins, Zone, Ornish, and LEARN diets for change in weight and related risk factors among overweight premenopausal women: the A TO Z Weight Loss Study: a randomized trial. JAMA. 2007 Mar 7;297(9):969-77. doi: 10.1001/jama.297.9.969. PMID 17341711
- [Background] Kossoff EH, Dorward JL. The modified Atkins diet. Epilepsia. 2008 Nov;49 Suppl 8:37-41. doi: 10.1111/j.1528-1167.2008.01831.x. PMID 19049584
- [Background] American Heart Association Nutrition Committee; Lichtenstein AH, Appel LJ, Brands M, Carnethon M, Daniels S, Franch HA, Franklin B, Kris-Etherton P, Harris WS, Howard B, Karanja N, Lefevre M, Rudel L, Sacks F, Van Horn L, Winston M, Wylie-Rosett J. Diet and lifestyle recommendations revision 2006: a scientific statement from the American Heart Association Nutrition Committee. Circulation. 2006 Jul 4;114(1):82-96. doi: 10.1161/CIRCULATIONAHA.106.176158. Epub 2006 Jun 19. PMID 16785338
- [Background] Law M. Dietary fat and adult diseases and the implications for childhood nutrition: an epidemiologic approach. Am J Clin Nutr. 2000 Nov;72(5 Suppl):1291S-1296S. doi: 10.1093/ajcn/72.5.1291s. PMID 11063471
- [Background] Mansoor N, Vinknes KJ, Veierod MB, Retterstol K. Effects of low-carbohydrate diets v. low-fat diets on body weight and cardiovascular risk factors: a meta-analysis of randomised controlled trials. Br J Nutr. 2016 Feb 14;115(3):466-79. doi: 10.1017/S0007114515004699. PMID 26768850
- [Background] Forsythe CE, Phinney SD, Fernandez ML, Quann EE, Wood RJ, Bibus DM, Kraemer WJ, Feinman RD, Volek JS. Comparison of low fat and low carbohydrate diets on circulating fatty acid composition and markers of inflammation. Lipids. 2008 Jan;43(1):65-77. doi: 10.1007/s11745-007-3132-7. Epub 2007 Nov 29. PMID 18046594
- [Background] Ness-Abramof R, Apovian CM. Waist circumference measurement in clinical practice. Nutr Clin Pract. 2008 Aug-Sep;23(4):397-404. doi: 10.1177/0884533608321700. PMID 18682591
- [Result] Lagiou P, Sandin S, Lof M, Trichopoulos D, Adami HO, Weiderpass E. Low carbohydrate-high protein diet and incidence of cardiovascular diseases in Swedish women: prospective cohort study. BMJ. 2012 Jun 26;344:e4026. doi: 10.1136/bmj.e4026. PMID 22735105
- [Result] Brehm BJ, Seeley RJ, Daniels SR, D'Alessio DA. A randomized trial comparing a very low carbohydrate diet and a calorie-restricted low fat diet on body weight and cardiovascular risk factors in healthy women. J Clin Endocrinol Metab. 2003 Apr;88(4):1617-23. doi: 10.1210/jc.2002-021480. PMID 12679447
- [Result] Yancy WS Jr, Olsen MK, Guyton JR, Bakst RP, Westman EC. A low-carbohydrate, ketogenic diet versus a low-fat diet to treat obesity and hyperlipidemia: a randomized, controlled trial. Ann Intern Med. 2004 May 18;140(10):769-77. doi: 10.7326/0003-4819-140-10-200405180-00006. PMID 15148063
- [Result] Organization WH. STEPS instruments for NCD risk factors (core and expanded version 1.4): the WHO STEPwise approach to Surveillance of noncommunicable diseases (STEPS). 2001
- [Result] Ervin RB. Prevalence of metabolic syndrome among adults 20 years of age and over, by sex, age, race and ethnicity, and body mass index: United States, 2003-2006. Natl Health Stat Report. 2009 May 5;(13):1-7. PMID 19634296
- [Result] Lakens D. Calculating and reporting effect sizes to facilitate cumulative science: a practical primer for t-tests and ANOVAs. Front Psychol. 2013 Nov 26;4:863. doi: 10.3389/fpsyg.2013.00863. PMID 24324449
- [Result] Brinkworth GD, Noakes M, Buckley JD, Keogh JB, Clifton PM. Long-term effects of a very-low-carbohydrate weight loss diet compared with an isocaloric low-fat diet after 12 mo. Am J Clin Nutr. 2009 Jul;90(1):23-32. doi: 10.3945/ajcn.2008.27326. Epub 2009 May 13. PMID 19439458
- [Result] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2985-3023. doi: 10.1016/j.jacc.2013.11.004. Epub 2013 Nov 12. No abstract available. PMID 24239920
- [Result] Krauss RM, Blanche PJ, Rawlings RS, Fernstrom HS, Williams PT. Separate effects of reduced carbohydrate intake and weight loss on atherogenic dyslipidemia. Am J Clin Nutr. 2006 May;83(5):1025-31; quiz 1205. doi: 10.1093/ajcn/83.5.1025. PMID 16685042
- [Result] Foster GD, Wyatt HR, Hill JO, Makris AP, Rosenbaum DL, Brill C, Stein RI, Mohammed BS, Miller B, Rader DJ, Zemel B, Wadden TA, Tenhave T, Newcomb CW, Klein S. Weight and metabolic outcomes after 2 years on a low-carbohydrate versus low-fat diet: a randomized trial. Ann Intern Med. 2010 Aug 3;153(3):147-57. doi: 10.7326/0003-4819-153-3-201008030-00005. PMID 20679559
- [Result] Rubins HB, Robins SJ, Collins D, Fye CL, Anderson JW, Elam MB, Faas FH, Linares E, Schaefer EJ, Schectman G, Wilt TJ, Wittes J. Gemfibrozil for the secondary prevention of coronary heart disease in men with low levels of high-density lipoprotein cholesterol. Veterans Affairs High-Density Lipoprotein Cholesterol Intervention Trial Study Group. N Engl J Med. 1999 Aug 5;341(6):410-8. doi: 10.1056/NEJM199908053410604. PMID 10438259
- [Derived] Ismael SA. Effects of low carbohydrate diet compared to low fat diet on reversing the metabolic syndrome, using NCEP ATP III criteria: a randomized clinical trial. BMC Nutr. 2021 Nov 3;7(1):62. doi: 10.1186/s40795-021-00466-8. PMID 34727975
- See also: STEPS Instrument for NCD Risk Factors (Core and Expanded Version 1.4) — https://apps.who.int